CLINICAL TRIAL: NCT04898686
Title: Study of the Probiotic Potential of a Lacticaseibacillus Strain in the Upper Airways in Patients With Allergic Rhinoconjunctivitis After Administration in a Chewable
Brief Title: Probiotic Chewables in Allergic Rhinoconjunctivitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Sarah Lebeer, Prof. dr.ir., University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B3002020000086
Record Dates: First submitted 2021-04-28; First posted 2021-05-24 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: lactobacilli; microbiome; probiotic chewables

STUDY DESIGN:
Intervention Model Description: double blind, randomized, placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): daily use of a probiotic chewable for 8 weeks
  Interventions: Biological: Probiotic chewables
- Placebo group (Placebo Comparator): daily use of the placebo chewable for 8 weeks
  Interventions: Biological: Placebo chewables

INTERVENTIONS:
Biological: Probiotic chewables — chewables containing Lacticaseibacillus rhamnosus GG
  Arms: Probiotic group
Biological: Placebo chewables — chewables without probiotic strain. Ingredients: Xylitol, microcrystalline cellulose, stearic acid, natural orange flavor, silica, magnesium stearate, citric acid and malic acid.
  Arms: Placebo group

SUMMARY:
With this double- blind, randomised, placebo-controlled study, the investigators want to investigate the influence of a chewable with the probiotic strain Lacticaseibacillus rhamnosus GG on the symptoms and immunological markers of allergic rhinoconjunctivitis (AR). In addition, the investigators aim to study the influence of this probiotic chewable on the microbiome of the upper respiratory tract after administration in adults with AR. The bacterial and cytokine profiles in the naso- and oropharynx will be monitored before, during and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 at the time of registration;
* Seasonal allergic rhinoconjunctivitis (AR) in the context of grass pollen allergy diagnosed on the basis of anamnesis cfr. ARIA guidelines and positive skin prick test and / or immunocap assay;
* Positive skin prick test (SPT) for grass pollen and / or the presence of specific IgE for grass pollen, confirmed by a medical specialist, measured at the start of the study: Soluprick SQ Phleum pratense pollen 10 HEP - ALK and / or IgE specific immunocap assay Phleum pratense (timothy grass) (g6);
* Body Mass Index in the range of 19-32 kg / m2;
* Instructed during screening and agreed not to use other probiotic products outside of the study during the study period;
* Signed the consent form.

Exclusion Criteria:

* Antibiotic use at baseline and during the study;
* Pregnant women;
* Unstable / uncontrolled asthma (to be determined by investigator-physician);
* Sensitization to dust mites
* History of probiotic use in the past two weeks;
* Current diagnosis of cancer or immunosuppressive therapy within the past 6 months;
* Abnormalities of the oral mucosa;
* Acute and chronic infectious and inflammatory upper airway diseases (eg acute / chronic rhinosinusitis cfr. EPOS guidelines);
* Clinically significant bleeding disorder;
* Any other medical condition that, in the principal investigator's opinion, warrants exclusion from the trial;
* History of regular use (> 3 days out of 7) of tobacco products within the previous two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Transfer of L. rhamnosus GG (estimated CFU counts) to the oronasopharyngeal cavity after administration of the chewable | at 8 weeks
  qPCR
Changes in the score of allergic rhinitis symptoms | over the study period (= 10 weeks)
  Daily questionnaires will be used, in which a self-reported Total Nasal Symptom Score (TNSS) based on rhinorrhea, nasal congestion, nasal itching and sneezing with symptom severity ranging from 0 (no problem) to 12 (very severe problem) will be recorded.

SECONDARY OUTCOMES:
changes in microbiome of the oronasopharyngeal region after administration of the chewable | baseline, 8 weeks
  16S rRNA amplicon sequencing
Inlfuence on general nose- and mouth health | baseline, 8 weeks, 10 weeks
  A clinical evaluation by an ENT specialist will be performed at the start and 8 weeks of the study to assess the general nose and mouth health of the participants. Questions on discomfort and symptoms of inflammation or infection in the nose and mouth will be included in the Sino-Nasal Outcome Test (SNOT-22)-based questionnaire implemented at the start, week 8 and week 10. Symptoms will be scored from 0 (no problem) to 5 (very severe problem)
Changes in the absolute numbers of specific airway pathogens and viruses | baseline, 8 weeks
  qPCR
Changes in cytokine levels (e.g. IL-10, IL-4, IL-5, IL-13) in oro- and nasopharynx samples, and cytokine and antibody levels in blood samples | baseline, 8 weeks
  qPCR and/or ELISA
Frequency of medication use | over the study period (= 10 weeks)
  Daily questionnaires will be used where the type and frequency of medication use should be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lebeer, Prof, Principal Investigator — Universiteit Antwerpen; Olivier Vanderveken, Prof, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Belgium